CLINICAL TRIAL: NCT00946348
Title: Cannabis and Schizophrenia: Self-Medication and Agonist Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Indiana University (Other); Columbia University (Other); University of Vermont (Other); University of Massachusetts, Worcester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: R01DA013196 (NIH); 1R01DA026799-01 (NIH); R01DA013196 (NIH); R01DA026799-01 (NIH); DPMC (Other: NIDA)
Record Dates: First submitted 2009-07-24; First posted 2009-07-27 (Estimated); Results first posted 2014-09-29 (Estimated); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: Schizophrenia; Dual Diagnosis; Schizoaffective Disorder; Psychotic Disorder; Cannabis Use Disorder
Keywords: Dronabinol; Schizophrenia; Dual Diagnosis; Substance Abuse; Cannabis Use Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Substance-Related Disorders | interventions — Dronabinol; nabiximols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dronabinol (Experimental): Dronabinol 10mg or 15 mg
  Interventions: Drug: Dronabinol
- Cannabis (Active Comparator): Cannabis cigarette
  Interventions: Drug: Cannabis

INTERVENTIONS:
Drug: Dronabinol — Dronabinol 10 mg or 15 mg
  Other Names: Marinol
  Arms: Dronabinol
Drug: Cannabis — Cannabis cigarette
  Other Names: Marijuana
  Arms: Cannabis

SUMMARY:
The first aim of this study is to determine whether a brain reward center (BRC) deficiency in patients with schizophrenia (SCZ) and cannabis use disorder (CUD) will be normalized when patients are given cannabis or dronabinol. The second aim will serve to further assess the effects of dronabinol on symptoms and medication side effects in this population.

DETAILED DESCRIPTION:
Cannabis use disorder (CUD) is up to ten times more common in schizophrenia (SCZ) than in the general population, and substantially worsens the course of this severe psychiatric disorder. Since SCZ occurs in 1% of the population, the comorbidity of CUD in 13% to 42% of people with this disorder presents society with an important public health problem. At present, treatments available for these "dual diagnosis" patients are inadequate. New treatments to limit cannabis use in patients with schizophrenia are sorely needed.

While the basis of substance use in patients with SCZ is not clear, some have suggested that use of substances may "self-medicate" negative symptoms or the side effects they experience from antipsychotic treatment. We have proposed an alternative formulation of this "self-medication hypothesis" -- a neurobiological formulation suggesting that a dysregulated mesocorticolimbic "brain reward circuit" (BRC) in patients with SCZ underpins their substance use, and that cannabis or other substance use ameliorates this dysregulated circuitry.

Our formulation is based on literature suggesting that the reinforcing effects of substances of abuse, including cannabis, may be related to their stimulation of dopamine (DA) neurons in the prefrontal cortex (PFC) and the mesolimbic system, key components of the BRC. Thus, according to this formulation, cannabis use "medicates" the dysregulated brain reward circuitry in patients with SCZ and allows them to have more normal responses to naturally rewarding events. Using a monetary probe linked to fMRI, we have demonstrated that patients with SCZ and co-occurring CUD (in agreement with preliminary studies from other investigators of non substance abusing patients) do indeed have a deficit within their BRC (reduced activation of the nucleus accumbens) as compared to normal subjects. This proposal will allow us to directly test the effects of cannabis on the BRC in patients with SCZ and CUD and thus to confirm our hypothesis regarding its effects in these patients. In addition, the proposal seeks to assess whether the cannabinoid agonist dronabinol, when given to patients with SCZ and CUD, will also ameliorate this BRC deficit, and, thus, whether dronabinol could be considered as a potential adjunctive treatment (given with an antipsychotic medication) to decrease their cannabis use.

The study will consist of two phases - a Pilot Study and the Main Study. The Pilot Study, completed in 10 "dual diagnosis" patients prior to the initiation of the Main Study, will establish the dose of oral dronabinol and the THC concentration of the cannabis cigarette to be used in the subsequent Main Study. The Main Study will involve 3 groups of subjects: two groups of dual diagnosis patients (with SCZ and co-occurring CUD), randomly assigned to one of the groups, and a group of healthy control patients. All subjects will be studied at baseline (T1) and 4 days later (T2) with a monetary probe linked to fMRI to evaluate their brain reward circuitry. At T1 all subjects will be tested without any intervention. At T2, patients in Groups 1 and 2 will receive both a dronabinol (or placebo) pill and a cannabis (or placebo cannabis) cigarette in a blinded fashion before testing. Group 1 patients will receive an active cannabis cigarette and a placebo pill; Group 2 patients will receive an active dronabinol pill and a placebo cannabis cigarette. Multiple measures will be taken to insure the safety of these patients during the use of cannabis and dronabinol. Group 3 (healthy controls) will not receive pill or cannabis cigarette and will serve as a control for repeated testing. Analyses will assess whether baseline BRC activation is different between patients and the control group, and whether use of cannabis and of dronabinol at T2 normalizes activation of BRC relative to T1 and relative to controls at T2.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for study subjects (dual diagnosis patients):

* Age 18-50;
* Diagnosis of schizophrenia or schizoaffective disorder (by SCID)
* Diagnosis of current cannabis abuse or dependence (by SCID);
* Recent use of cannabis (within the past month on Timeline Follow-Back);
* Stability on antipsychotic medication for past 1 month);
* Outpatient status for past 3 months;
* Willing and able to participate as demonstrated by a signed informed consent document.

Inclusion criteria for normal control subjects:

* Age 18-50;
* Willing to participate as demonstrated by a signed informed consent document

Exclusion Criteria:

Exclusion criteria for study subjects (dual diagnosis patients):

* PANSS subscale for positive symptoms of psychosis item > 3 [moderate] on Day 15 (once they are abstinent from cannabis);
* Cocaine/stimulant use disorder;
* Pharmacological treatment for addiction (e.g., disulfiram, naltrexone, acamprosate, topiramate); Mental retardation;
* Pregnancy or currently nursing;
* Uncontrolled serious medical condition;
* Seizure disorder
* Seeking treatment to limit their cannabis use
* Taking clozapine

Additional Exclusion criteria for Main Study patients only:

* Claustrophobia prohibiting scanning
* History of head injury with period of unconsciousness;
* Metal objects within the body;
* Taking antipsychotic other than risperidone or first generation antipsychotic as main treatment
* Previous participation in the Pilot Dose Finding Study

Exclusion criteria for normal control subjects:

* Axis I or Axis II psychiatric diagnosis (including substance use disorder) based on SCID
* Mental retardation;
* History of head injury with period of unconsciousness;
* Metal objects within the body;
* Pregnancy or currently nursing;
* Uncontrolled serious medical condition;
* Current tobacco smokers. Note: We exclude current tobacco smoking (but not a history of smoking) in the normal control subjects since the fact of cigarette smoking could select subjects with a dysregulated BRC as a basis for their continued cigarette smoking in the face of social conventions toward non-smoking.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2009-12; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan I Green, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was conducted through Dartmouth Hitchcock Medical Center, and local community mental health centers.
Pre-assignment Details: Of the 52 people who consented to participate in the study, 12 met eligibility criteria for the main study and were randomized. Because persons who met entry criteria received study treatment on only one day, all randomized participants completed the study.
Groups:
- Dronabinol: Dronabinol 15 mg
- Cannabis: Cannabis cigarette (3.6% THC)
Period: Overall Study
Arm/Group | Dronabinol | Cannabis
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 52 subjects consented; 15 were in a pilot study to determine the dose of dronabinol and strength of the marijuana cigarette and 14 were health controls (who received no drug)for comparison. The remaining 23 subjects consented to the Main Study and 12 were met eligibility criteria and were randomized to receive dronabinol or a marijuana cigarette.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dronabinol | Cannabis | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 12
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.17 (8.32) | 36.2 (9.6) | 34.2 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: fMRI Connectivity of Regions of Interest (ROI) Within the Brain Reward Circuitry (BRC).
Description: Average Z scores for the region-of-interest functional connectivity at the second scan (when subjects received either a cannabis cigarette or 15mg of dronabinol) between the bilateral nucleus accumbens (NAc) and ventral anterior cingulate cortex (vACC) for patients with schizophrenia and co-occurring cannabis use disorder.
Time Frame: Measures were acquired at peak THC level for each of the two drugs up to 4 hours.
Measure: Mean (Standard Deviation); unit: Z score
Arm/Group | Dronabinol | Cannabis
Number analyzed (Participants) | 6 | 6
Z score | .40 (.85) | .33 (.38)

2. Secondary Outcome: To Assess the Effects of Dronabinol in This Population to Determine Whether Measures of Craving, Mood and Negative Symptoms Will Improve Using the PANSS; and to Determine Whether Measures of Psychotic Symptoms and Cognitive Deficits Will Increase.
Time Frame: Over 8 hours
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from the date of consent through the final telephone contact with the patient after the second scan. Though the time differed based on scheduling of patients, it was typically 4-5 weeks.
Arm/Group | Dronabinol | Cannabis
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 2/6 | 3/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dronabinol (N=6) | Cannabis (N=6)
Cannabis Withdrawal (Psychiatric disorders) | 2 (5) | 3 (11) — This was assessed using the Cannabis Withdrawal Assessment Scale at each visit. On any day that a participant scored greater than 12, he or she would be considered to be experiencing cannabis withdrawal.
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Increased Psychiatric Symptoms (Psychiatric disorders) | 0 (0) | 1 (1) — The actual symptom that increased was not noted but was believed to be secondary to cannabis withdrawal.
Decreased Sleep (Psychiatric disorders) | 1 (1) | 0 (0)
Less Appetite (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No